CLINICAL TRIAL: NCT05541783
Title: A Multi-center Prospective Randomized Controlled Trial Comparing the Quality of Life Between Laparoscopic-assisted Distal Gastrectomy (LADG) and Totally Laparoscopic Distal Gastrectomy (TLDG) for Gastric Cancer
Brief Title: Laparoscopic-assisted Distal Gastrectomy and Totally Laparoscopic Distal Gastrectomy for Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, PHD,MD, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LATDG
Record Dates: First submitted 2022-09-06; First posted 2022-09-15 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer，Laparoscopic distal gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laparoscopy-assisted distal gastrectomy (Active Comparator): The patients who are assigned to LADG group undergo extracorporeal anasto- mosis for gastrointestinal reconstruction.
  Interventions: Procedure: laparoscopy-assisted distal gastrectomy Group
- Totally laparoscopic distal gastrectomy (Experimental): The patients who are allocated to TLDG group undergo intracorporeal anastomosis for the recovery of gastrointes- tinal continuity after gastrectomy.
  Interventions: Procedure: Totally laparoscopic distal gastrectomy

INTERVENTIONS:
Procedure: laparoscopy-assisted distal gastrectomy Group — LADG
  Arms: Laparoscopy-assisted distal gastrectomy
Procedure: Totally laparoscopic distal gastrectomy — TLDG
  Arms: Totally laparoscopic distal gastrectomy

SUMMARY:
The aim of this study is comparing the short-term quality of life between laparoscopy-assisted distal gastrectomy and totally laparoscopic distal gastrectomy for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20-80 years;
2. Patients had an Eastern Cooperative Oncology Group performance status score of 0 or 1;
3. Patients had histologically confirmed gastric adenocarcinoma (tumor size<5cm) at clinical stage I-III with T1-4aN0-2M0 excluding T4b or N3 tumors, according to the of the American Joint Committee on Cancer classification system, eighth edition;
4. Patients were expected to undergo laparoscopic distal gastrectomy with D2 lymphadenectomy.

Exclusion Criteria:

1. Patients had bulky regional lymph nodes (larger than 3 cm at the long diameter) or possible distant metastasis in preoperative evaluation
2. Patients had history of chemotherapy, radiotherapy, immunotherapy or target therapy;
3. Patients had any concurrent or previous malignant tumor;
4. Patients had unstable cardiovascular, respiratory, kidney, or liver disease and poorly controlled hypertension, diabetes, mental disorders; history of upper abdominal surgery (except laparoscopic cholecystectomy).
5. Patients were histologically proven gastric adenocarcinoma (by preoperative gastrofiberscopy).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Scores on the physical function and pain symptom scales of EORTC QLQ-C30 questionnaire | 30 days postoperatively
  Scores on the physical function and pain symptom scales of EORTC QLQ-C30 questionnaire at 30 days postoperatively

SECONDARY OUTCOMES:
Scores on the other scales of EORTC QLQ-C30 questionnaire postoperatively | 30 days postoperatively
  Scores on the other scales of EORTC QLQ-C30 questionnaire at 30 days postoperatively
Scores on EORTC QLQ-C30 questionnaire | 7 days and 90 days postoperatively
  Scores on EORTC QLQ-C30 questionnaire at 7 days and 90 days postoperatively
Scores on the scales of EORTC QLQ-STO22 questionnaire postoperatively | 7，30 and 90 days postoperatively
  Scores on the scales of EORTC QLQ-STO22 questionnaire at 7，30 and 90 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Dazhi Xu, PHD, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No